CLINICAL TRIAL: NCT04034225
Title: An Open-Label, Multi-Center Trial of SNS-301 Added to Pembrolizumab in Patients With Locally Advanced Unresectable or Metastatic/Recurrent Squamous Cell Carcinoma of the Head and Neck
Brief Title: Addition of SNS-301 to Checkpoint Inhibitor Treatment in Metastatic/Recurrent SCCHN
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated by the sponsor
Sponsor: Sensei Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNS-301-2-2
Record Dates: First submitted 2019-07-16; First posted 2019-07-26 (Actual); Results first posted 2022-12-30 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SNS-301 added to pembrolizumab (Experimental): * SNS-301
  * Pembrolizumab
  Interventions: Drug: SNS-301; Drug: Pembrolizumab

INTERVENTIONS:
Drug: SNS-301 — Day 0, Week 3, Week 6, Week 9 then every 6 weeks (±3 days) for 6 additional doses, thereafter every 12 weeks (±3 days) up to 24 months.
Drug: Pembrolizumab — Pembrolizumab (200 mg dose) IV infusion will be administered over 30 minutes every 3 weeks up to 24 months or Pembrolizumab (400 mg dose) IV will be administered over 30 minutes every 6 weeks up to 24 months.
  Other Names: Keytruda

SUMMARY:
To evaluate safety, immunogenicity and anti-tumor responses of intradermally delivered SNS-301 added to checkpoint inhibitor therapy in locally advanced unresectable or metastatic/recurrent squamous cell carcinoma of the head and neck (SCCHN) patients.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, multi-center trial to evaluate the safety, immunogenicity and preliminary clinical efficacy of SNS-301 delivered intradermally in addition to pembrolizumab in patients with locally advanced unresectable or metastatic/recurrent SCCHN. The trial population consists of patients with locally advanced unresectable or metastatic/recurrent SCCHN who are currently receiving checkpoint inhibitor (CPI) therapy (Cohort A) or are naïve to CPI therapy (Cohort B). Patients who are currently receiving CPI therapy must have a best response of stable disease (SD) or first evidence of progressive disease (PD) after a minimum of 12 weeks of treatment with a CPI. Patients receiving a CPI other than pembrolizumab will be switched over to pembrolizumab at the time of entering this study. Patients receiving pembrolizumab in the first line setting must be PD-L1 positive.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Be 18 years of age or older.
3. Have histologically or cytologically documented locally advanced unresectable or metastatic/recurrent SCCHN and meet the criteria of either Cohort A or B.

   Cohort A: Patients with Ongoing CPI Therapy
   1. Patients currently receiving a checkpoint inhibitor (CPI: anti-PD-1 and anti-PD-L1 agents).
   2. Patients currently receiving a CPI must be considered by Investigator to have the potential to derive clinical benefit from continued treatment with pembrolizumab.
   3. Based on RECIST 1.1/iRECIST criteria on current CPI treatment (prior to initiation of this study), patients must have a best response of stable disease (SD) or first evidence of progressive disease (PD) after a minimum of 12 weeks of a CPI.
   4. Patients on other CPI therapy than pembrolizumab must be willing to switch over to pembrolizumab therapy.

   Cohort B: Patients without Previous CPI Therapy
   1. Patients must be checkpoint inhibitor naïve (anti-PD-1 and anti-PD-L1 agents)
   2. Patients should receive study treatment as first line (PD-L1 positive) or as second line (PD-L1 negative) systemic therapy in the advanced/metastatic setting.
4. Have measurable disease by RECIST 1.1.
5. Eastern Cooperative Oncology Group (ECOG) Performance Scale 0-1.
6. Have a life expectancy of ≥ 3 months.
7. Be willing to provide a pre-treatment tissue sample (archived or fresh).
8. Demonstrate adequate organ function: hematological, renal, hepatic, coagulation parameters.
9. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use two highly effective contraceptive methods during the treatment period and for at least 180 days after the last dose of study treatment. For male patients: Agree that during the period specified above, men will not father a child. Male patients must remain abstinent, must be surgically sterile during the treatment period and for at least 180 days after the last dose of study treatment.

Exclusion Criteria:

1. Any approved anti-cancer therapy including chemotherapy, targeted small molecule therapy or radiation therapy within 2 weeks prior to trial Day 0.
2. Participated on a clinical trial of an investigational agent and/or investigational device within 28 days prior to Day 0.
3. Uncontrolled tumor-related pain.
4. Malignancies other than indications open for enrollment within 3 years prior to Day 0.
5. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
6. Known hypersensitivity allergy or contraindication to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the PD-1/PD-L1 inhibitor formulation.
7. Active autoimmune disease that has required systemic treatment in the past 2 years
8. History or any evidence of interstitial lung disease.
9. History of HIV. HIV antibody testing recommended per investigator's clinical suspicion.
10. Active hepatitis B (hepatitis B surface antigen reactive) or active hepatitis C (HCV qualitative RNA detected); testing recommended per investigator's clinical suspicion.
11. Severe infections within 4 weeks prior to enrollment.
12. Received therapeutic oral or IV antibiotics within 2 weeks prior to Day 0.
13. History or current evidence of any condition, therapy or laboratory abnormality that in the opinion of the treating investigator might confound the results of the trial.
14. Prior allogeneic stem cell or solid organ transplant.
15. Known previous or ongoing, active psychiatric or substance abuse disorders that would interfere with the requirements of the trial.
16. Treatment with systemic immunomodulating agents (including but not limited to IFNs, IL-2, ipilimumab) within 6 weeks or five half-lives of the drug, whichever is shorter, prior to first dose.
17. Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi Melhem, MD, Study Director — Sensei Biotherapeutics
Locations (10):
- United States (10):
  - University of California - San Francisco, San Francisco, California
  - Christiana Care, Newark, Delaware
  - Georgetown University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - Alliance for Multispeciality Research, Kansas City, Missouri
  - Mt. Sinai, New York, New York
  - New Orleans Clinical Research, Knoxville, Tennessee
  - Clear Lake Specialties, Webster, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in the article, after deidentification (text, tables, figures and appendices) will be shared to researchers who have provide a methodologically sound proposal and sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Access will be considered to researchers who provide a methodologically sound proposal. Analysis must achieve the aims outlined in the approved proposal Proposals should be directed to info@senseibio.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 36 months following article publication.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were required to provide archival biopsy material or have a fresh biopsy prior to dosing.
Groups:
- SNS-301 Added to Pembrolizumab: * SNS-301
  * Pembrolizumab
  SNS-301: Day 0, Week 3, Week 6, Week 9 then every 6 weeks (±3 days) for 6 additional doses, thereafter every 12 weeks (±3 days) up to 24 months.
  Pembrolizumab: Pembrolizumab (200 mg dose) IV infusion will be administered over 30 minutes every 3 weeks up to 24 months or Pembrolizumab (400 mg dose) IV will be administered over 30 minutes every 6 weeks up to 24 months.
Period: Overall Study
Arm/Group | SNS-301 Added to Pembrolizumab
Started | 25 (Study stopped prematurely. 25/60 patients enrolled.)
Completed | 0
Not Completed | 25
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2
Not completed — Study termination by Sponsor | 18
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Groups:
- SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD; SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy: * SNS-301
  * Pembrolizumab
  SNS-301: Day 0, Week 3, Week 6, Week 9 then every 6 weeks (±3 days) for 6 additional doses, thereafter every 12 weeks (±3 days) up to 24 months.
  Pembrolizumab: Pembrolizumab (200 mg dose) IV infusion will be administered over 30 minutes every 3 weeks up to 24 months or Pembrolizumab (400 mg dose) IV will be administered over 30 minutes every 6 weeks up to 24 months.
- Total: Total of all reporting groups
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy | Total
Number analyzed (Participants) | 21 | 4 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (7.42) | 53.3 (13.10) | 61.1 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 17 | 3 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 4 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 2 | 18
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 4 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events of SNS-301 in Addition to Pembrolizumab
Description: Number of adverse events including adverse events of special interest as assessed by CTCAE v5.0
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 21 | 4
Participants | 16 | 3

2. Primary Outcome: Objective Response Rate by RECIST and iRECIST
Description: Objective response rate based on best objective response during the study. Objective tumor response definitions included: Complete response (CR): Disappearance of all target lesions, Partial response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters, Progressive disease (PD): At least a 20% increase in the sum of diameters of the target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm and Stable disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 18 | 1
Participants
  Partial Response | 1 | 0
  Stable Disease | 8 | 1
  Progressive Disease | 9 | 0

3. Primary Outcome: Duration of Response by RECIST 1.1 and iRECIST
Description: Duration of response calculated from date of first response to date of progression. Objective tumor response definitions included: Complete response (CR): Disappearance of all target lesions, Partial response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters, Progressive disease (PD): At least a 20% increase in the sum of diameters of the target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm and Stable disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study.
Time Frame: 12 weeks
Population: A total of 18 patients were evaluable in patients who had previous pembrolizumab group and 1 patient was evaluable in the CPI naive group. One patient had a partial response with a DOR of 48.3 weeks. All other patients had stable disease or has progressive disease at the 12 week timeframe.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 18 | 1
weeks | 48.3 [NA to NA] — only 1 participant with a partial response which was 48.3 weeks. | 0 [NA to NA] — no participants met the criteria for efficacy.

4. Primary Outcome: Disease Control Rate by RECIST 1.1 and iRECIST
Description: Disease control rate calculated as the proportion of patients with stable disease or better. Objective tumor response definitions included: Complete response (CR): Disappearance of all target lesions, Partial response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters, Progressive disease (PD): At least a 20% increase in the sum of diameters of the target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm and Stable disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 18 | 1
participants | 9 | 1

5. Primary Outcome: Progression Free Survival by RECIST 1.1 and iRECIST
Description: Progression free survival calculated from the date of start of treatment to date of progression. Objective tumor response definitions included: Complete response (CR): Disappearance of all target lesions, Partial response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters, Progressive disease (PD): At least a 20% increase in the sum of diameters of the target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm and Stable disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study.
Time Frame: 12 weeks
Population: 19/25 patients were evaluable for this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 18 | 1
Participants | 9 | 1

6. Primary Outcome: Overall Survival
Description: Overall survival calculated from date of treatment to date of death.
Time Frame: 36 months
Population: Study stopped prematurely; no patients were assessed at 36 months thus no data collected. At the time of termination, four deaths occurred in the patients previously receiving pembrolizumab group and no deaths in the CPI naive group.
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Antigen-specific Response
Description: Measure levels at pretreatment, changes during treatment and at progression or end of study
Time Frame: 12 weeks
Population: 16/25 patients were evaluable for this assessment.
Measure: Number; unit: ASPH antigen-specific responders
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 15 | 1
ASPH antigen-specific responders | 0 | 0

8. Secondary Outcome: TCR Sequencing
Description: Determine TCR diversity pretreatment, changes during treatment and at progression or end of study
Time Frame: 12 weeks
Population: Blood samples were collected. However, due to the lack of ASPH-specific T-cell responses in patients treated with SNS-301 and the subsequent discontinuation of the clinical trial, the samples were not analyzed and no data were generated.
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Immune Gene Transcript Profiling
Description: Determine gene signature pretreatment, during treatment and at progression
Time Frame: 12 weeks
Population: as for outcome 8
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Profiling of Pro-inflammatory/Immunosuppressive Molecules
Description: Measure levels at pretreatment, changes during treatment and at progression or end of study
Time Frame: 12 weeks
Population: as for outcome 8
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Immune Related Expression
Description: Determine immune expression pretreatment, changes during treatment and at progression
Time Frame: 12 weeks
Population: as for outcome 8
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Tumor Specific Oncoproteins
Description: Determine expression pretreatment, during treatment and at progression
Time Frame: 12 weeks
Population: as for outcome 8
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: ASPH Expression
Description: Determine pretreatment expression, changes during treatment and at progression
Time Frame: 12 weeks
Population: as for outcome 8
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Cytokine/Chemokine Profiling
Description: Determine cytokine/chemokine profile pretreatment, changes during treatment and at progression
Time Frame: 12 weeks
Population: as for outcome 8
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: ctDNA
Description: Determine ctDNA profile pretreatment, changes during treatment and at progression
Time Frame: 12 weeks
Population: as for outcome 8
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from study entry through 30 days post the patient's last dose. On average, patients were on the study for 3.3 months.
Description: AE definition as per clinicaltrials.gov definition
Arm/Group | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy
All-Cause Mortality (participants affected / at risk) | 3/21 | 0/4
Serious Adverse Events (participants affected / at risk) | 5/21 | 1/4
Other Adverse Events (participants affected / at risk) | 16/21 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD (N=21) | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy (N=4)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SNS-301 Added to Pembrolizumab in Participants on a CPI >12 Weeks With a BOR SD/uPD (N=21) | SNS-301 Added to Pembrolizumab in Participants CPI Naive/ First Line Systemic Therapy (N=4)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0)
Injection site discomfort (General disorders) | 1 (1) | 0 (0)
Mass (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Secretion discharge (General disorders) | 1 (1) | 0 (0)
Swelling face (General disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 0 (0)
White blood cell count increased (Investigations) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolongation (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study stopped prematurely for lack of efficacy 25 patients were enrolled. Lab analyzes were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Submission of data for publication/presentation will be reviewed, coordinated and approved by Sensei in collaboration with the Investigator.

DOCUMENTS (2):
  • Study Protocol (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT04034225/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT04034225/SAP_001.pdf